CLINICAL TRIAL: NCT01609153
Title: A Randomized Double-blind Controlled Trial to Assess the Benefits of Olanzapine and Amisulpride Combination Treatment in Acutely Ill Schizophrenia Patients. - COMBINE
Brief Title: Comparison of Antipsychotic Combination Treatment of Olanzapine and Amisulpride to Monotherapy
Acronym: COMBINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMBINE
Record Dates: First submitted 2012-05-23; First posted 2012-05-31 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; amisulpride; olanzapine; polypharmacy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Amisulpride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Olanzapine or Placebo (Active Comparator)
  Interventions: Drug: Amisulpride; Drug: Olanzapine and Amisulpride
- Amisulpride or Placebo (Active Comparator)
  Interventions: Drug: Olanzapine; Drug: Olanzapine and Amisulpride
- Olanzapine and Amisulpride (Active Comparator)
  Interventions: Drug: Olanzapine; Drug: Amisulpride

INTERVENTIONS:
Drug: Olanzapine — Coated tablet 5-20 mg milligram(s) per day for 16 weeks
  Other Names: Zyprexa
  Arms: Amisulpride or Placebo; Olanzapine and Amisulpride
Drug: Amisulpride — 200-800 mg milligram(s)per day for 16 weeks
  Other Names: Amisulprid Hexal
  Arms: Olanzapine and Amisulpride; Olanzapine or Placebo
Drug: Olanzapine and Amisulpride — Zyprexa:
  Coated tablet 5-20 mg milligram(s) per day for 16 weeks
  Amisulpride:
  Coated tablet 200-800 mg milligram(s)per day for 16 weeks
  Other Names: Zyprexa, Amisuprid Hexal
  Arms: Amisulpride or Placebo; Olanzapine or Placebo

SUMMARY:
A study to examine whether an antipsychotic combination treatment of olanzapine and amisulpride is more effective than olanzapine and amisulpride alone.

DETAILED DESCRIPTION:
Polypharmacy in antipsychotic therapy is an important issue when treating patients with schizophrenia. It is not well confirmed that a combination of two antipsychotic drugs lead to therapeutic benefit in contrast to monotherapy. However there is a highly frequent practice of combining atypical non-clozapine treatment that could be due to potential benefits when seeking alternatives to a high rate of non-response in acute phase. Therefore there is a need for further trials of sufficient power to address efficacy and safety issues of this regimen. Combining two selected atypical drugs in a complementary way may minimize side-effects and enhance efficacy. In order to specify these advantages it is intend to examine approaches to combination treatment: Amisulpride and olanzapine show complementing receptor binding profiles and have shown to have efficacy and good tolerability when administered in combination in retrospective studies. The object of this trial is to study whether acutely ill patients with combination of amisulpride and olanzapine are more frequently in symptomatic remission after 8 weeks than those with olanzapine or amisulpride monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia and schizoaffective disorder according to International Classification of Diseases (ICD-10);
* age 18-65;
* Positive and Negative Symptom Scale Total-Score ≥ 70 and two items of the positive symptom subscale ≥4.
* voluntary treatment after written informed consent
* legal capacity
* exclusion of pregnancy by laboratory test (Beta HCG)

Exclusion Criteria:

* participation in other interventional studies with drugs or medical devices
* first episode patients
* physical disease that might have effects on the conduct or evaluation of the trial
* contraindications to medication according to experts information
* oversensitivity to active substance or other component of the drugs used
* known clozapine resistance
* suicidal ideation
* pregnancy or lactation
* which of pregnancy or absence save contraception
* dependency to sponsor or investigator
* institutionalization through judicial or regulatory order
* oversensitivity to placebo (mannite/aerosil)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement of schizophrenia after 8 weeks of treatment in comparison to time of inclusion of patient measured py Positive and Negative Symptom Scale (PANSS) | 8 weeks
  Whether there is a symptomatic improvement of schizophrenia after 8 weeks of treatment in comparison to time of inclusion of patient measured py Positive and Negative Symptom Scale (PANSS)

SECONDARY OUTCOMES:
Symptomatic improvement of schizophrenia after 16 weeks of treatment in comparison to time of inclusion of patient measured py PANSS total score reduction | 16 weeks.
  To study whether a combination treatment of olanzapine and amisulpride show a PANSS total score reduction from baseline to week 16.
Symptomatic improvement of schizophrenia from baseline to week 2 up to week 16 measured by PANSS total score reduction. | Every 2 weeks up to week 16.
  Whether a combination treatment of olanzapine and amisulpride show a PANSS total score reduction from baseline to every 2 weeks up to week 16.
PANSS total score reduction from baseline to week 2 as a predictor of the change after 8 weeks | 8 weeks
  Whether a change of PANSS total score reduction from baseline to week 2 is a predictor of the change after 8 weeks
Serious adverse drug reactions | 16 weeks
  Frequency and severity of serious adverse drug reactions
Change of clinical condition measured by Clinical Global Impression Scale (CGI scale) | every 2 weeks from baseline up to week 16
  Whether there is a change of clinical condition measured by Clinical Global Impression Scale (CGI scale)
Change of the subjective well-being measured by Subjective Wellbeing under Neuroleptics Scale (SWN-K) | between week 0, 8, 16
  Whether there is a change of the subjective well-being measured by Subjective Wellbeing under Neuroleptics Scale(SWN-K)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schmidt-Kraepelin, Dr., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (21):
- Germany (21):
  - RWTH Aachen, Aachen
  - Rheinhessen Fachklinik Alzey, Alzey
  - Rhein-Mosel-Fachklinik Andernach, Andernach
  - Bezirkskliniken Schwaben, Bezirkskrankenhaus Augsburg, Augsburg
  - Charite-Universitätsmedizin Berlin, Berlin
  - LVR-Klinikum Köln, Cologne
  - LWL-Klinik Dortmund, Dortmund
  - LVR-Klinikum Düsseldorf, Düsseldorf
  - Universitätsmedizin Göttingen, Göttingen
  - Zentrum für Seelische Gesundheit Kreiskliniken Darmstadt-Dieburg Standort: Groß-Umstadt, Groß-Umstadt
  - Klinik für Psychiatrie, Psychotherapie und Psychosomatik am Bezirkskrankehaus Günzburg, Günzburg
  - Klinik für Psychiatrie, Sozialpsychiatrie und Psychotherapie Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - LVR-Klinik Langenfeld, Langenfeld
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Leipzig
  - Universitätsmedizin Mainz Klinik für Psychiatrie und Psychotherapie, Mainz
  - Zentralinstitut für Seelische Gesundheit, Mannheim
  - LMU München, München
  - TU München, München
  - Bezirksklinikum Regensburg, Klinik für Psychiatrie und Psychotherapie, Regensburg
  - Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Derived] Schmidt-Kraepelin C, Feyerabend S, Engelke C, Riesbeck M, Meisenzahl-Lechner E, Verde PE, Correll CU, Kluge M, Makiol C, Neff A, Lange C, Englisch S, Zink M, Langguth B, Poeppl TB, Reske D, Gouzoulis-Mayfrank E, Grunder G, Hasan A, Brockhaus-Dumke A, Jager M, Baumgartner J, Leucht S, Cordes J; COMBINE Study Group. Amisulpride and olanzapine combination treatment versus each monotherapy in acutely ill patients with schizophrenia in Germany (COMBINE): a double-blind randomised controlled trial. Lancet Psychiatry. 2022 Apr;9(4):291-306. doi: 10.1016/S2215-0366(22)00032-3. Epub 2022 Mar 8. PMID 35276079